CLINICAL TRIAL: NCT01006031
Title: Efficacy of High Doses of Both Pegylated Interferon Alfa-2a and Ribavirin for Retreatment of HIV-coinfected Patients With Liver Cirrhosis Due to HCV Genotype 1 or 4 Nonresponders to Previous Standard Therapy.
Brief Title: Retreatment With High Doses of pegIFN Alfa-2a and Ribavirin of Previous Nonresponders HIV-coinfected Patients With Cirrhosis Due to HCV 1-4
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sociedad Andaluza de Enfermedades Infecciosas (Network)
Responsible Party: Principal Investigator, Antonio Rivero, Luis Fernando Lopez-Cortes, Sociedad Andaluza de Enfermedades Infecciosas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEPAVIR_IFN_2009
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Liver Cirrhosis; Hepatitis C Virus; HIV Infection
Keywords: Liver cirrhosis; Hepatitis C virus; HIV infection; Pegylated interferon alfa-2a; Ribavirin; Treatment experienced
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C; HIV Infections | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PegIFN alfa-2a and Ribavirin (Experimental): HIV-coinfected patients with compensated cirrhosis by hepatitis C virus, genotype 1 or 4.
  Interventions: Drug: Pegylated interferon alfa-2a and Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a and Ribavirin — Pegylated interferon alfa-2a (360 ug per week) plus oral Ribavirin (800 mg b.i.d.) for 48 or 72 weeks. The treatment will be discontinued for patients who did not achieve a reduction with respect to baseline of at least 0.5 log10 IU/ml in plasma RNA-HCV levels at week 4 or 2 log10 UI/ml at week 12 and will be considered as viral failures.
  Duration: 48 weeks for patients reaching an undetectable plasma RNA_HCV at week12 and 72 weeks for those without a negative viremia at week 12 but a reduction of at least 2 log10 IU/ml in RNA-HCV levels.
  Other Names: Pegasys; Copegus

SUMMARY:
Objective: To evaluate the efficacy and safety of high doses of both peginterferon-alfa 2a (360 ug per week) plus ribavirin (800 mg b.i.d.) in HIV-infected patients with compensated liver cirrhosis by HCV genotype 1 or 4 without previous virological response(*) to a standard dose treatment of both drugs.

(*) Non previous virological response: no decrease of plasma RNA-HCV at least 2 log10 after 12 weeks in treatment or breakthrough viremia while on treatment.

Additionally, this study will evaluated the influence of simultaneous peginterferon-alfa 2a and ribavirin plasma concentrations on early viral response (EVR) and sustained viral response (SVR) in these patients.

Method: Pilot clinical trial, phase II-III, open labeled multicenter in which patients from several hospitals of the Servicio Andaluz de Salud will be enrolled.

The usual clinical and analytical follow up will be performed but additional blood samples will be obtained for determination of interferon and ribavirin plasma levels. The primary end point will be a sustained virologic response (defined as an undetectable serum HCV-RNA after 24 weeks after the cessation of treatment). Likewise, rapid virological response (at 4 weeks of treatment), early virological response (at 12 weeks), and end of treatment response rates will be evaluated as well as their relationships with the plasma interferon an ribavirin concentrations determined by ELISA and HPLC, respectively. The safety and tolerability of the studied medications will be evaluated by means of clinical adverse events, physical examination and laboratory results. The evolution of liver fibrosis will be evaluated comparing the basal and end of treatment results of transient elastometry.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* HIV-infected patients with compensated liver cirrhosis by HCV genotype 1 or 4 without previous virological response(*) to a standard dose treatment of both drugs.
* Women of child-bearing age: negative pregnancy test
* Ability to understand and sign a written consent form

Exclusion Criteria:

* HCV genotypes different to 1 or 4
* Acute or chronic hepatitis B infection (positivity for hepatitis B surface antigen or plasma DNA) or other concomitant causes of liver disease
* Pregnancy or breast feeding.
* Decompensated liver disease at baseline.
* Neutropenia <1000/uL, anemia <100 g/L or thrombocytopenia <20.000/uL.
* Creatinine clearance < 50 mL/min.
* Concomitant treatment with immunomodulators or zidovudine, didanosine or stavudine.
* Organ or bone marrow transplantation
* Current alcoholism or iv drug abuse. Methadone is allowed.
* Current neoplasm and/or anti-tumor chemotherapy or immunomodulators
* Psychosis or uncontrolled clinical depression
* Auto-immune disease, including auto-immune hepatitis
* History of significant cardiovascular disease (NYHA III-IV) including but not limited to uncontrolled hypertension, angina pectoris, myocardial infarction, coronary artery surgery and congestive heart failure.
* Thyroid dysfunction.
* Clinically significant retinal abnormalities
* Inability to understand and sign a written consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Sustained viral response (undetectable serum HCV-RNA) | Throughout treatment and 24 weeks after finishing it

SECONDARY OUTCOMES:
Relationships between the plasma interferon an ribavirin concentrations and efficacy | Throughout treatment and 24 weeks after finishing it.
safety and tolerability of the studied medications | Throughout treatment and 24 weeks after finishing it
The evolution of liver fibrosis will be evaluated comparing the basal and end of treatment results of transient elastometry | baseline and after finishing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Lopez-Cortes, MD, PhD, Study Director — Instituto de Biomedicina de Sevilla. Hospitales Universitarios Virgen del Rocío; Luis F Lopez-Cortes, MD, PhD, Principal Investigator — Instituto de Biomedicina de Sevilla. Hospitales Universitarios Virgen del Rocio; Antonio Rivero, MD, PhD, Principal Investigator — Hospital Universitario Reina Sofia. Cordoba; Mª Jose Rios-Villegas, MD, PhD, Principal Investigator — Hospital Universitario Viren MAcarena. Sevilla; Juan A. Pineda, MD, PhD, Principal Investigator — Hospital Universitario de Valme. Sevilla
Locations (4):
- Spain (4):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospitales Universitarios Virgen del Rocío, Seviila
  - Hospital Universitario de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville